CLINICAL TRIAL: NCT04781608
Title: In It Together: Using Acceptance and Commitment Therapy to Treat Distress Among Older Adults With Sensory Loss and Their Spouses
Acronym: SoS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Velux Fonden (Other)
Responsible Party: Principal Investigator, Camilla Stine Øverup, Postdoc, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VELUX 22361; 1779339 (Other: Danish Data Protections Agency); 504-0225/20-5000 (Other: University of Copenhagen Research Ethics Committee for Science and Health)
Record Dates: First submitted 2021-01-18; First posted 2021-03-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Sensory Loss (Impairment of Sight and/or Hearing)
Keywords: Sensory loss; Hearing impairment; Sight impairment; Elderly couples; Age 60 or older; Online; Digital; Intervention; Acceptance and Commitment therapy
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions: 1) Intervention group, which will receive access to the digital intervention program, and 2) Control group, who will not receive immediate acess to the digital intervention program.
  Intervention group:
  Participants will be asked to complete survey measures at baseline (prior to access to the 4-module digital intervention program), 6-weeks, 10 weeks, and 18 weeks.
  Control group:
  Participants will be asked to complete survey measures at baseline , 6-weeks, and 10 weeks (control group participants gain access to the digital intervention program after completion of the 10-week survey).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Gains access to the digital intervention program
  Interventions: Behavioral: English: In It Together (IIT)
- Wait-list- control group (No Intervention): Does not gain access to the intervention (until end of study)

INTERVENTIONS:
Behavioral: English: In It Together (IIT) — Digital intervention program that consists of 4 modules, to be completed 1 week apart. The modules consist of psychoeducation, as well as acceptance and commitment therapy-inspired activities.
  Other Names: Danish: Sammen on Sansetab (SOS)
  Arms: Intervention group

SUMMARY:
Impairments in hearing and/or vision are common in older age. Having lived one's life as a fully sighted and hearing individual, older adults with sensory loss must come to terms with their declining capacity to interact with others and waning independence. There is ample research evidence showing that sensory loss (i.e., loss of hearing, vision or both) can be a distressful experience for older adults and their spouses, yet little has been done to understand what works in alleviating this distress or develop scalable cost-effective interventions to counter this distress or associated outcomes like depression, anxiety, poor quality of life, and lower relationship quality. In this project, the investigators will design and test an easy-to-administer, online intervention aimed at reducing emotional and marital distress in older adults with sensory loss and their spouses. The goal of the intervention will be to develop acceptance of the sensory loss through a series of Acceptance and Commitment Therapy inspired educational, self-compassion, and therapeutic activities. In prior research, acceptance has been flagged as a promising factor on which to intervene to assist older couples' emotional and marital recovery in the context of sensory loss. Thus, the investigators expect that the intervention should show encouraging results regarding the alleviation of distress in this group and contribute significantly to the psychosocial rehabilitation of older adults with sensory loss and their spouses.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years of age or older
* Be able to read and write in Danish
* Be in a romantic relationship of at least 1 year
* Live together with the partner (share housing)
* Feel either one self or one's partner has a sensory loss (hearing and/or sight) that affects day-to-day life. This sensory loss does not need to be confirmed by a health care provider.

Exclusion Criteria:

* Less than 60 years of age
* Cannot read or write in Danish
* Not in a romantic relationship
* Relationship length of less than 1 year
* Not living together with the partner (not share housing)
* Currently receiving psychological help (therapy/intervention)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
WHO-5 well-being | Within the last 2 weeks
  5-item measure of general well-being (Bech, 1999, 2012)
Couple Satisfaction Index | Follow-up 1: During the last 6 weeks
  4-item measure of satisfaction with one's romantic relationship (Funk & Rogge, 2007)
Depression | Within the last 2 weeks
  9-item measure of depressive symptoms (PHQ-9; Kroenke, Spitzer, & Williams, 2001; Kroenke
  & Spitzer, 2002)

SECONDARY OUTCOMES:
Psychological flexibility | Follow-up 1: During the last 6 weeks
  7-item measure of psychological flexibility (AAC-II; Bond, Hayes, Baer, Carpenter, Guenole, Orcutt, Waltz, & Zettle, 2011).
Communication | Follow-up 1: During the last 6 weeks
  12-item measure of satisfaction with communication with partner (Jones, Jones, & Morris, .018)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla S Øverup, PhD, Principal Investigator — University of Copenhagen; Gert Martin Hald, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We will share all individual data, along with a data dictionary and analytic code. The data will be anonymized prior to sharing. The materials will be uploaded to a data repository (which as yet to be determined)
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will be shared after June 30th, 2022.